CLINICAL TRIAL: NCT04303546
Title: VOPITB a New Devices to Determine Peripheral Arterial Stiffness: Protocol for Validation Study
Brief Title: VOPITB a New Devices to Determine Peripheral Arterial Stiffness: Validation Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Sergio Rico Martín, PhD. RN. Associate Professor, University of Extremadura
Other Study IDs: VOPITB STUDY
Record Dates: First submitted 2020-03-08; First posted 2020-03-11 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Cardiovascular Risk Factor; Cardiovascular Diseases; Atherosclerosis of Artery
Keywords: arterial stiffnes; pulse wave velocity; VOPITB; validation
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- < 30 years
  Interventions: Device: arterial stiffness measurements
- 30-60 years
  Interventions: Device: arterial stiffness measurements
- > 60 years
  Interventions: Device: arterial stiffness measurements

INTERVENTIONS:
Device: arterial stiffness measurements — We will measure arterial stiffness by VOPITB and with others devices to validate VOPITB

SUMMARY:
Our group has developed a device called "Velocidad Onda de Pulso Indice Tobillo Brazo (VOPITB)" . In this device the oscillometric method is used for easily and accurately measure the pulse wave velocity PWV in the arms and legs separately, allowing new arterial stiffness indices to be studied (sum, difference, ratio, baPWV and CAVI). The aim of our study will be to validate the PWV measures by VOPITB with other references devices that measures arterial stiffness. Moreover we will perform a clinical study to assess the clinical utility of VOPITB.

ELIGIBILITY:
Inclusion Criteria:

* Subjects ≥ 18 years who agree to participate in the study and do not meet any of the exclusion criteria.

Exclusion Criteria:

* History of CVD (ischaemic heart disease, stroke or peripheral arterial disease)
* Atrial fibrillation or other cardiac rhythm disorders
* Pacemaker-dependent
* Impalpable arterial pulse at site of measurement
* Pregnancy
* Terminal condition
* Age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The sample size has been calculated in order to provide that a difference between the CAVI values obtained from measurement of both devices, VOPITB and VaSera, shall be up to of 0.8 points in comparison with the CAVI reference values for Spanish adults population [21]. the base parameters used to calculate the sample size were as follows: standard deviation (sd) of CAVI measured by VaSera VS-1500 and VOPITB (1.44), mean difference between CAVI measurements (0.8), confidence level (95%), and power (80%). Thus, the estimated sample size was found as 102 patients. In addition, for compensating possible incomplete data sets from patients who could withdraw or fail to complete the study, 20% were added. Finally, a total of 120 subjects (a minimum of 40% of subjects for each gender group) will be evaluated according to the following criteria:
  * < 30 years (40 subjects)
  * 30 - 60 years (40 subjects)
  * > 60 years (40 subjects)
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-03-08 (Estimated); Primary Completion 2020-04-15 (Estimated); Study Completion 2020-12-15 (Estimated)

PRIMARY OUTCOMES:
cardio-ankle vascular index (CAVI) validation | 8 months
  We will determine CAVI with VOPITB, as well as its validation against the reference device (VaSera VS-1500) and assess its clinical utility.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rico Martin S, Vassilenko V, de Nicolas Jimenez JM, Rey Sanchez P, Serrano A, Martinez Alvarez M, Calderon Garcia JF, Sanchez Munoz-Torrero JF. Cardio-ankle vascular index (CAVI) measured by a new device: protocol for a validation study. BMJ Open. 2020 Oct 20;10(10):e038581. doi: 10.1136/bmjopen-2020-038581. PMID 33082193